CLINICAL TRIAL: NCT05715684
Title: Patient-Centered Surgical Prehabilitation
Acronym: Prehab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Principal Investigator, Matthew Mossanen, MD, Urologic Surgeon, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-329
Record Dates: First submitted 2023-01-18; First posted 2023-02-08 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Bladder Cancer; Cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard treatment Plan (Other): This is the main arm of the study in which all 25 anticipated participants will be enrolled into.
  Interventions: Other: Exercise Training; Dietary Supplement: Nutritional Intervention

INTERVENTIONS:
Other: Exercise Training — Virtually supervised exercise training for four weeks prior to cystectomy
Dietary Supplement: Nutritional Intervention — Patients scheduled to undergo cystectomy will receive liquid Ensure supplemental shakes for 2 weeks prior to surgery and liquid Ensure supplemental shakes for 1 week postoperatively

SUMMARY:
The purpose of this research is to validate the prehabilitation program which is defined as a set of interventions meant to prepare the body physically and nutritionally for the cystectomy procedure.

DETAILED DESCRIPTION:
This research study is testing the efficacy of the prehabilitation study which is a set of investigational interventions and also tries to define the most appropriate and effective set type of interventions to use for further studies. "Investigational" means that the intervention is being studied. In this research study, the investigators hope to learn whether or not this combination of prehabilitation interventions has an impact on the recoverability of participants who will undergo cystectomy or bladder removal surgery. The 5 interventions that make up the prehabilitation study are:

* Participant Interview (If one of the first ten participants)
* Exercise Testing
* Exercise Training
* Nutritional Support
* Clinical Assessment of Nutritional Status

ELIGIBILITY:
Inclusion Criteria:

1. Patents must be candidates for all types of cystectomy surgery including urinary diversion via open or robotic approach.
2. Patients between the ages 18 and 85 years
3. American Society of Anesthesiologists (ASA) Physical Status Score of class 1-4
4. Ileal conduit or ileal neobladder urinary diversion
5. Able to understand the study procedures, agreed to participate in the study program, and voluntarily provided informed consent

Exclusion Criteria:

1. Scheduled for a partial cystectomy
2. Previous total colectomy, gastrectomy, or gastric bypass, or functional colostomy or ileostomy
3. More than three doses of opioids (oral or parenteral) within 7 days before the day of surgery
4. The presence of metastatic cancer
5. Be undergoing treatment for another type of cancer concurrently
6. Chemotherapy for bladder cancer within 1 month of scheduled surgery; prior neoadjuvant chemotherapy allowed.
7. Pregnant (identified by a positive serum pregnancy test administered after the initial screening process and before the commencement of study activities) or lactating, or not postmenopausal (no menses for at least 1 year) and of childbearing potential and not using an accepted method of birth control (i.e, surgical sterilization; intrauterine contraceptive device; oral contraceptive, diaphragm, or condom in combination with contraceptive cream, jelly, or foam; or abstinence) (Participants will be asked to use birth control for the entire study and for at least 2 weeks after the last dose of study drug.)
8. Participated in another investigational drug or medical device study within 30 days of surgery or planning to be enrolled in another investigational drug or medical device study or any study in which active patient participation was required outside normal hospital data collection during the course of this study
9. Clinically significant laboratory abnormalities at screening that would have resulted in the cancellation of surgery
10. Using illicit drugs or abusing alcohol
11. History of previous surgeries, illness, or behavior (eg, depression, psychosis) that in the opinion of the investigator might have confounded the study results or might have posed additional risk in administering the study procedures
12. Patients with severe dementia (as determined from medical records and history. Severe dementia will be defined as dementia that impacts daily functioning.)
13. Patients with severe hepatic impairment as defined by Child-Pugh Class C. Patients with Child-Pugh Class A-B hepatic impairment are eligible for the study.
14. A history of heart failure.
15. Patients with end-stage renal disease as defined by GFR <15.
16. Patients with heart failure.
17. Patients with complete gastrointestinal obstruction.
18. Patients with gastrostomy tube, jejunostomy tube or who require enteral tube feeds.
19. Non-English-speaking patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-12-27 (Estimated); Study Completion 2027-12-25 (Estimated)

PRIMARY OUTCOMES:
Total days hospitalized within 30-days of surgery | 60 months
  This is the total number of days within 30 days after bladder removal surgery, that a patient is hospitalized.
Length of stay | 60 months
  This is the total length of stay in days after bladder removal surgery
Number and type of minor and major complications | 60 months
  This is the number and types of major and minor complications which occur post bladder removal surgery
Discharge disposition | 60 months
  This is the disposition of the patient at discharge or when the patient is released from the hospital.
Readmissions | 60 months
  This is the number of times a patient that was discharged come back to the hospital for any issue related to their bladder removal surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation